CLINICAL TRIAL: NCT00438217
Title: Analysis of Genetic and Environmental Parameters Influencing Growth Rate of Precocious Puberty Children
Acronym: CPP-EDG 01
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Pisa (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CPP-EDG 01
Record Dates: First submitted 2007-02-21; First posted 2007-02-22 (Estimated); Last update posted 2007-02-22 (Estimated); Status verified 2007-02

CONDITIONS: Central Precocious Puberty
Keywords: precocious puberty, genetics, environmental factors
MeSH Terms: conditions — Puberty, Precocious | interventions — Triptorelin Pamoate; Leuprolide

INTERVENTIONS:
Drug: Triptorelin (GnRH agonists)
Drug: Leuprolide (GnRH agonists)

SUMMARY:
The goal of CPP-EDG 01 study is to assess possible genetic and/or environmental parameters which may influence the growth rate of children affected by precocious puberty. In this view, we are collecting clinical data and biological samples of children attended as outpatients at the Pediatric Endocrine Center of Pisa from 1998 to present (the study is still open). From biological (blood) samples, gene polymorphisms such as endocrine disruptor levels are determined and compared to different growth pattern of pediatric patients treated with different GnRH agonists.

ELIGIBILITY:
Inclusion Criteria:

* Clinica diagnosis of central precocious puberty
* Diagnosis is based on growth spurt, bone age advancement, positive GnRH agonist stimulating test, pubertal sex steroid levels before 8 years of age for female and 9 years for male, respectively

Exclusion Criteria:

* Thyroid disorders
* Peripheric diagnosis of precocious puberty
* Genetic disorders

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 100

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Saggese, MD, Study Director — Department of Pediatrics, University of Pisa
Locations (1):
- Center of Pediatric endocrinology, Department of Pediatrics, University of Pisa, Pisa, Italy